CLINICAL TRIAL: NCT00479076
Title: A Single Agent-combination Hybrid Phase I, Open-label, Dose-escalation Study of the Safety, Tolerability, and Pharmacokinetics of Intravenous AVE0005 (VEGF Trap)Administered Every 2 Weeks in Combination With Oral S-1 in Patients With Advanced Solid Malignancies
Brief Title: A Phase I Study of Intravenous Aflibercept in Combination With S-1 in Japanese Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TED10089
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Neoplasms
Keywords: antineoplastic agents; VEGF Trap
MeSH Terms: conditions — Neoplasms | interventions — aflibercept; S 1 (combination)

INTERVENTIONS:
Drug: aflibercept (AVE0005) — intravenous infusion
Drug: S-1 — oral administration

SUMMARY:
The primary objective of this study is to determine the recommended phase II dose of AVE0005 in combination with S-1 in Japanese cancer patients.

The secondary objectives of this study are to assess the safety profile of AVE0005, to determine the pharmacokinetics of AVE0005, to make a preliminary assessment of antitumor effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer patients without standard of care
* ECOG performance status 0, 1, or 2
* Adequate organ and bone marrow function

Exclusion Criteria:

* Need for a major surgery or radiation therapy during the study
* History of hypersensitivity to S-1
* Known dihydropyrimidine dehydrogenase deficiency
* Uncontrolled hypertension
* History of brain metastases
* Ascites requiring drainage
* Pregnancy or breastfeeding
* Patients who have previously been treated with AVE0005

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2007-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) defined as grade 3 or higher National Cancer Institute - Common Terminology Criteria (NCI-CTC) toxicities | during the first cycle of study treatment

SECONDARY OUTCOMES:
safety: physical examination, laboratory safety tests, adverse events | treatment period
pharmacokinetic values | treatment period
objective response rate | treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Tokyo, Japan